CLINICAL TRIAL: NCT05598476
Title: Effect of Chest Compression on Respiratory Mechanics in ARDS Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2022PI154
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 5kg bag — a 5 kg bag is applied on the chest for 2 hours

SUMMARY:
In some ARDS patients, a mild chest compression (5 kg) improves lung compliance.

We aim to determine wether such an improvement is due to a better recruitment or to a reduction of overdistension

ELIGIBILITY:
Inclusion Criteria:

* ARDS (Berlin definition)
* Age >18y
* under invasive mechanical ventilation

Exclusion Criteria:

* people protected by the law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ARDS patients under invasive mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
respiratory mechanics | 2 hours

IPD SHARING:
Plan to Share IPD: No